CLINICAL TRIAL: NCT07085650
Title: The Multi-center Study of Comprehensive Atrial Fibrillation Regurgitation by 3-dimensional Transoesophageal Echocardiography and Recurrent Events Evaluation
Brief Title: The Multi-center Study of Comprehensive Atrial Fibrillation Regurgitation and Recurrent Events Evaluation
Status: Recruiting | Type: Observational
Sponsor: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Chunyan Ma, Professor, First Hospital of China Medical University
Other Study IDs: CARE-AF STUDY
Record Dates: First submitted 2024-12-18; First posted 2025-07-25 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-05

CONDITIONS: Atrial Fibrillation (AF); Mitral Regurgitation; Tricuspid Regurgitation
MeSH Terms: conditions — Atrial Fibrillation; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- AF group

SUMMARY:
Atrial fibrillation (AF) is the most common cardiac arrhythmia in the clinic and can lead to valve regurgitation and a poor prognosis. At present, atrial fibrillation ablation is one of the most effective means for the recurrence of atrial fibrillation in clinical practice, but the recurrence rate is high. Therefore, it is of great significance to find the predictors of relapse after atrial fibrillation ablation for clinical precision treatment. three-dimensional transesophageal ultrasound (3D-TEE) can comprehensively evaluate the valve regurgitation, flap ring changes, atrial or auricular thrombosis in patients with atrial fibrillation. It is also a necessary examination before atrial fibrillation ablation.

Therefore, this study intends to combine 3D-TEE and three-dimensional transthoracic echocardiographic (3D-TTE) examination to evaluate the cardiac structure and function of patients. To comprehensively evaluate atrial fibrillation valve regurgitation and explore the predictors of recurrence after atrial fibrillation ablation.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia in clinical practice. It is characterized by disturbance of atrial electromechanical activity, and the incidence rate of the general population can reach 1.5-2%. Valvular regurgitation may be associated with atrial fibrillation, leading to poor prognosis. However, due to limited screening techniques, it is difficult to comprehensively evaluate valvular regurgitation and its influencing factors. On the other hand, AF may lead to reduced heart function, atrial or auricular thrombosis, and lead to high risk events such as ischemic stroke and heart failure.

Therefore, restoring normal sinus rhythm is of great significance for patients with atrial fibrillation. Atrial fibrillation ablation is one of the most effective methods for atrial fibrillation reversion, which is of great significance for improving the prognosis of patients. However, although the current ablation is very mature and effective, the recurrence rate one year after the first ablation can reach 20 to 40%. The high recurrence rate not only increases the readmission risk of patients and increases the economic burden, but also makes some patients shy away from ablation therapy and delay treatment, resulting in adverse outcomes. At present, there is a lack of effective indicators for predicting the recurrence of atrial fibrillation after ablation in clinical practice. Therefore, it is of great significance to search for predictive factors for the recurrence of atrial fibrillation after ablation in clinical precision treatment.

three-dimensional transesophageal ultrasound (3D-TEE) can comprehensively evaluate the valve regurgitation, flap ring changes, atrial or auricular thrombosis in patients with atrial fibrillation. It is also a necessary examination before atrial fibrillation ablation.

Therefore, this study intends to combine 3D-TEE and three-dimensional transthoracic echocardiographic (3D-TTE) examination to evaluate the cardiac structure and function of patients. To comprehensively evaluate atrial fibrillation valve regurgitation and explore the predictors of recurrence after atrial fibrillation ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old;
2. Patients who came to the hospital with atrial fibrillation and intended to undergo ablation.

Exclusion Criteria:

1. - History of left atrial or left atrial appendix thrombus, new cerebral infarction and myocardial infarction (< 6 months);
2. Congenital heart disease, valvular heart disease, dilated heart disease, hypertrophic cardiomyopathy, pacemaker implantation, artificial valve replacement;
3. hyperthyroidism, severe liver and kidney insufficiency;
4. Proposed cardiac pacemaker implantation;
5. Previous history of catheter ablation;
6. The quality of three-dimensional transesophageal images was insufficient and could not be analyzed;
7. refuse to sign the informed consent.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation population in China
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial fibrillation | 3 months after atrial fibrillation ablation
  Using 12-lead electrocardiogram and 24h-holter electrocardiogram to exam patients. The recurrence of atrial fibrillation is defined as atrial tachycardia, atrial flutter or atrial fibrillation lasting for 30 seconds or more.

OTHER OUTCOMES:
mitral or tricuspid regurgitation improvement | 3 months after atrial fibrillation ablation
  1. Utilize three-dimensional ultrasound technology to measure multiple parameters of the mitral valve annulus and tricuspid valve annulus, including annulus area (cm2), circumference (cm), non-planar angle (°), etc. Compare the differences of these parameters with the baseline state at 3 months.
  2. Use Doppler technology to assess the improvement or deterioration of mitral and tricuspid regurgitation, including regurgitation diameter (mm), regurgitation area (cm2).

CONTACTS AND LOCATIONS:
Locations (1):
- First Hospital of China Medical University, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No